CLINICAL TRIAL: NCT00001335
Title: New Therapeutic Strategies for Patients With Ewing's Sarcoma Family of Tumors, High Risk Rhabdomyosarcoma, and Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930125; 93-C-0125
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Ewing's Sarcoma; Neuroblastoma; Rhabdomyosarcoma
Keywords: Peripheral Stem Cell Transfusion; Up-Front Phase II Window; Dose-Intensive Vincristine; Dose-Intensive Doxorubicin; Dose-Intensive Cyclophosphamide; ADR-529 for Cardioprotection; BID Radiation Therapy for Local Control
MeSH Terms: conditions — Sarcoma, Ewing; Neuroblastoma; Rhabdomyosarcoma | interventions — Dexrazoxane; Topotecan; Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: ADR-529
Drug: Topotecan
Drug: G-CSF

SUMMARY:
The prognosis for patients with metastatic Ewing's sarcoma family of tumors (ESF), rhabdomyosarcoma (RMS), and neuroblastoma (NBL) remains dismal, with less than 25% long-term disease-free survival. Though less grave, the prognosis for cure for other high-risk patients is approximately 50%. New treatment strategies, including the identification of highly active new agents, maximizing the dose intensity of the most active standard drugs, and the development of improved methods of consolidation to eradicate microscopic residual disease, are clearly needed to improve the outcome of these patients. This protocol will address these issues by commencing with a Phase II window, for the highest risk patients, to evaluate a series of promising drugs with novel mechanisms of action. All patients will then receive 5 cycles of dose-intensive "best standard therapy" with doxorubicin (adriamycin), vincristine, and cyclophosphamide (VAdriaC). Patients at high risk of relapse will continue onto a phase I consolidation regimen consisting of three cycles of dose-escalated Melphalan, Ifosfamide, Mesna, and Etoposide (MIME). Peripheral blood stem cell transfusions (PBSCT) and recombinant human G-CSF will be used as supportive care measures to allow maximal dose-escalation of this combination regimen.

DETAILED DESCRIPTION:
The prognosis for patients with metastatic Ewing's sarcoma family of tumors (ESF), rhabdomyosarcoma (RMS), and neuroblastoma (NBL) remains dismal, with less than 25% long-term disease-free survival. Though less grave, the prognosis for cure for other high-risk patients is approximately 50%. New treatment strategies, including the identification of highly active new agents, maximizing the dose intensity of the most active standard drugs, and the development of improved methods of consolidation to eradicate microscopic residual disease, are clearly needed to improve the outcome of these patients. This protocol will address these issues by commencing with a Phase II window, for the highest risk patients, to evaluate a series of promising drugs with novel mechanisms of action. All patients will then receive 5 cycles of dose-intensive "best standard therapy" with doxorubicin (adriamycin), vincristine, and cyclophosphamide (VAdriaC). Patients at high risk of relapse will continue onto a phase I consolidation regimen consisting of three cycles of dose-escalated Melphalan, Ifosfamide, Mesna, and Etoposide (MIME). Peripheral blood stem cell transfusions (PBSCT) and recombinant human G-CSF will be used as supportive care measures to allow maximal dose-escalation of this combination regimen.

ELIGIBILITY:
The patient must fall into one of the following diagnostic categories:

Ewing's sarcoma family of tumors (ESF): Includes Ewing's sarcoma (classic, atypical, extra-osseous), primitive sarcoma of bone, ectomesenchymoma, or peripheral primitive neuroectodermal tumor (peripheral neuroepithelioma).

Rhabdomyosarcoma: The patient must have either

High-risk arm: Metastatic disease at diagnosis (any site, any histology);

OR

Moderate-risk arm: Incompletely resected ( Clinical Group III) Stage II tumors and ALL stage III tumors (regardless of degree of surgical resection).

Neuroblastoma: Any patient with metastatic disease at diagnosis (POG stage D or Evans' stage IV); or, patients with loco-regional metastatic disease (POG stage C) or tumor infiltrating across the midline (Evans' stage III) IF they have an elevated serum ferritin (greater than 142 ng/ml), an amplified N-myc copy number (greater than 10 copies on Southern analysis), or a DNA index of greater than 1.1.

The patient must not have been previously treated with chemotherapy or radiation therapy.

Patients must be greater than or equal to 1 year of age but less than or equal to 25 years of age. Patients weight must be greater than or equal to 15 kg.

The patient (or his/her guardian if less than 18 years of age) must sign a document indicating that he/she is aware of the investigational nature of this treatment protocol and the potential risks and benefits that may be expected.

Potentially fertile female patients must have a documented negative urine or serum pregnancy test.

Patients must have a documented negative HIV serologic evaluation (Western Blot and/or ELISA).

Patients must not have abnormal cardiac function (left ventricular ejection fraction less than 45% as measured by gated equilibrium radionuclide angiography [MUGA scan] and confirmed by echocardiography).

Patients must not have impaired renal function (serum creatinine greater than or equal to twice the upper limit of normal for age).

Patients with a total bilirubin of greater than 4.0 mg/dl (or a direct bilirubin of greater than 2.0 mg/dl) or SGOT/SGPT greater than five times the upper limits of normal (NOT on the basis of hepatic involvement by tumor) will be excluded.

Patients with a second malignancy following previous therapy will be excluded.

Patients previously treated with chemotherapy or radiation therapy (other than limited, emergency radiation therapy) will be excluded.

Patients who are HIV-infected will be excluced.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1993-04; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States